CLINICAL TRIAL: NCT01534065
Title: A Multi-center, Post Marketing Surveillance Study to Monitor the Safety and Performance of the Barricaid® ARD in the Treatment of Back and Radicular Pain Caused by Primary Lumbar Disc Herniation
Brief Title: Barricaid EU Post Market Study for Primary Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BARD-CP-001
Record Dates: First submitted 2012-01-04; First posted 2012-02-16 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Lumbar Disc Herniation
Keywords: Hernia; Intervertebral Disk Displacement; Pathological Conditions, Anatomical; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia; Pathological Conditions, Anatomical; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Barricaid (Experimental): CE Marked Device
  Interventions: Device: Barricaid

INTERVENTIONS:
Device: Barricaid — Implanted intra-operatively during discectomy

SUMMARY:
The purpose of this multi-center post marketing surveillance study is to monitor the safety and performance of the Barricaid® ARD when used to surgically reconstruct the anulus of the L1 - S1 spinal disc.

DETAILED DESCRIPTION:
The purpose of this prospective, randomized, multicenter study is to demonstrate the superiority of the Barricaid® when used as an adjunct to a primary lumbar limited discectomy (as described by Spengler), to limited discectomy alone, with regard to preventing reherniation and the recurrence of pain or dysfunction. Patients, ages 21 - 75, will have, in part, a positive straight leg raise (or positive femoral stretch, as appropriate), MRI confirmation of a disc herniation, and minimum Oswestry and VAS leg scores of 40 out of 100 to qualify for this study. Additional patient criteria can be found in the inclusion/exclusion criteria section.

Superiority of the Barricaid relative to limited discectomy alone will be based on a comparison of overall success rates of the Barricaid and a concurrent group (randomized) of control patients treated by primary lumbar limited discectomy at select European (approximately 15-20) sites.

This study has two co-primary endpoints. Success of the study will be based on the Barricaid population achieving statistical superiority over the concurrently randomized non-implanted limited discectomy population at 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (male or female).
2. Patients with posterior or posterolateral disc herniations at one or two levels between L1 and S1 with radiographic confirmation of neural compression using CT and/or MRI.
3. At least six (6) weeks of failed, conservative treatment prior to surgery, including physical therapy, use of anti-inflammatory medications at maximum specified dosage and/or administration of epidural/facet injections.;
4. Minimum posterior disc height of 3mm at the index level(s).
5. Lower back pain and/or sciatica with or without spinal claudication.
6. Oswestry Questionnaire score of at least 40/100 at baseline.
7. VAS leg pain of at least 40/100 at baseline.

Exclusion Criteria:

1. Spondylolisthesis Grade II or higher
2. Subject requires uni or bilateral facetectomy to treat leg/back pain
3. Subject has back or non-radicular leg pain of unknown etiology.
4. Prior fusion (with or without instrumentation), motion preservation, facetectomy or IDET surgery at the index lumbar vertebral level
5. Subject's requiring a spine DEXA (i.e., patients with SCORE of ≥ 6) with a T Score less than -2.0 at the index level.
6. Subject has clinically compromised vertebral bodies at the index level(s) due to any traumatic, neoplastic, metabolic, or infectious pathology.
7. Subject has sustained pathologic fractures of the vertebra or multiple fractures of the vertebra or hip.
8. Subject has scoliosis of greater than ten (10) degrees (both angular and rotational).
9. Any metabolic disease bone disease that has not been stabilized for at least three months (e.g., Paget's disease, osteomalacia, osteogenesis imperfecta, thyroid and/or parathyroid gland disorder, etc.).
10. Subject has an active infection either systemic or local.
11. Subject has cauda equine syndrome or neurogenic bowel/bladder dysfunction.
12. Subject has severe arterial insufficiency of the legs (Screening on physical examination= patients with diminution or absence of dorsalis pedis or posterior tibialis pulses. If diminished or absent by palpation, then an arterial ultrasound is required with vascular plethysmography. If the absolute arterial pressure is below 50mm of Hg at the calf or ankle level, then the patient is to be excluded) or other peripheral vascular disease).
13. Subject has significant peripheral neuropathy, patient defined as a patient with Type I or Type II diabetes or similar systemic metabolic condition causing decreased sensation in a stocking-like or non-radicular and non-dermatomal distribution in the lower extremities.
14. Subject has insulin-dependent diabetes mellitus.
15. Subject is morbidly obese (defined as a body mass index >40, or weighs more than 100 lbs over ideal body weight).
16. Subject has been diagnosed with active hepatitis, AIDS, or HIV.
17. Subject has been diagnosed with rheumatoid arthritis or other autoimmune disease.
18. Subject has a known allergy to titanium, polyethylene or polyester materials.
19. Subject is pregnant or interested in becoming pregnant in the next three (3) years.
20. Subject has active tuberculosis or has had tuberculosis in the past three (3) years.
21. Subject has a history of active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no signs or symptoms of the malignancy for at least two (2) years.
22. Subject is immunologically suppressed, received steroids >1 month over the past year.
23. Currently taking anticoagulants, other than aspirin, unless the patient can be taken off the anticoagulant for surgery
24. Subject has a current chemical/alcohol dependency or significant psychosocial disturbance.
25. Subject has a life expectancy of less than three (3) years.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Patient function as measured on Oswestry Disability Index (ODI) | 24 months
  15-point reduction in ODI at 24-month visit relative to baseline
Disc height maintenance as measured from standing x-rays | 24 months
  75% maintenance at 2 years relative to pre-op, measured by independent radiologist, (reference: Yorimitsu, et al, Spine 2001)
Clinically symptomatic recurrent herniation at the index level, confirmed by imaging | 24 months
  Performed at 24 months by the Investigator.
Migration of the bone anchor posteriorly into the epidural space | 24 months
  Radiographic imaging taken to ensure no migration of the device. Assessment made by the Investigator and Radiographic Core lab.
Removal or revision of the implant | 24 months
  Any removal or revision of the implant will be measured as a safety outcome.
Supplemental fixation applied at the treated level | 24 months
  Any supplemental fixation applied at the treated level will be tracked.

SECONDARY OUTCOMES:
Back Pain on Visual Analog Scale (VAS) | 24 months
  Back pain on VAS will be tracked.
Leg Pain on Visual Analog Scale (VAS) | 24 months
  Leg pain assessment will be tracked. Patient reported outcome.
Quality of life on SF36 | 24 months
  Quality of life on SF36 will be tracked. Patient reported outcome.
Comparison of neurological symptoms on clinical examination, relative to baseline | 24 months
  Patient will have the following examinations: straight leg raising, deep tendon reflexes, forward bend, motor strength examination (hip flexors, knee extensors, tibialis, long toe extensors), and sensory (light touch, pin prick, or vibration)
Frequency of AE's | 24 months
  Frequency of AE's reported throughout the study will be tracked and analyzed at the 24 month visit.

CONTACTS AND LOCATIONS:
Overall Officials: Claudius Thome, PhD, Principal Investigator — University of Innsbruck, Department of Neurosurgery

REFERENCES:
- [Result] Lequin MB, Barth M, Thome C, Bouma GJ. Primary limited lumbar discectomy with an annulus closure device: one-year clinical and radiographic results from a prospective, multi-center study. Korean J Spine. 2012 Dec;9(4):340-7. doi: 10.14245/kjs.2012.9.4.340. Epub 2012 Dec 31. PMID 25983843
- [Result] Bouma GJ, Barth M, Ledic D, Vilendecic M. The high-risk discectomy patient: prevention of reherniation in patients with large anular defects using an anular closure device. Eur Spine J. 2013 May;22(5):1030-6. doi: 10.1007/s00586-013-2656-1. Epub 2013 Feb 3. PMID 23377540